CLINICAL TRIAL: NCT01330004
Title: The Relationship of Systolic and Diastolic Blood Pressure Changes Over Time to Patient Outcomes in Incident Hemodialysis Patients
Brief Title: Blood Pressure Change and Outcome
Acronym: BP
Status: Completed | Type: Observational
Sponsor: Renal Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 080-11
Record Dates: First submitted 2011-03-31; First posted 2011-04-06 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Renal Disease; High Blood Pressure
MeSH Terms: conditions — Kidney Diseases; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hemodialysis patients

SUMMARY:
Hyper- and hypotension are important predictors of survival in non-ESRD (end stage renal disease) population. In dialysis patients, however, it has been shown that higher blood pressure levels may actually be beneficial to patient outcomes. Dynamics of blood pressure evolution over time has not been previously studied in dialysis population. The investigators aim to understand how both blood pressure levels and blood pressure changes over time predict patient survival.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal Research Institute hemodialysis patients
Sampling Method: Non-Probability Sample
Enrollment: 12695 (Actual)
Dates: Start 1999-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Effect size of the relation of dynamic changes of blood pressure (BP) at different ranges of BP to survival in incident hemodialysis patients. | Up to 11 years and 11 months
  The ranges of blood pressure measurements in mmHg over time and the relation to patient outcomes (including survival)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan W Levin, MD, Principal Investigator — Renal Research Institute
Locations (1):
- Renal Research Institute, New York, New York, United States

REFERENCES:
- [Derived] Raimann JG, Usvyat LA, Thijssen S, Kotanko P, Rogus J, Lacson E Jr, Levin NW. Blood pressure stability in hemodialysis patients confers a survival advantage: results from a large retrospective cohort study. Kidney Int. 2012 Mar;81(6):548-58. doi: 10.1038/ki.2011.426. Epub 2012 Jan 4. PMID 22217879